CLINICAL TRIAL: NCT03161925
Title: Chinese Liver Cancer Clinical Survey
Acronym: CLCS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Insight Science & Technology Co. Ltd. (Other)
Responsible Party: Sponsor
Other Study IDs: INW161116CLCS
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Primary Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to make better use of clinical resources of the real world, strengthen the standardization of PLC diagnosis and treatment, and constantly improve the academic level of liver cancer in China, we intends to launch "Chinese Liver Cancer clinical Survey" project in cancer specialized hospitals and large general hospitals and to explore the best clinical pathway of PLC multidisciplinary consultation.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) is one of the most common malignant tumors of digestive system and also a serious threat to the health and safety of Chinese people, and has caused serious economic burden to the country. Research purposes: To understand the clinical characteristics of patients with primary liver cancer (PLC) in China; To investigate the etiology and pathogenesis of PLC in China; To understand the current status of clinical treatment of PLC in China, and to analyze the gaps among these conditions and domestic treatment guidelines, industry consensus, the international treatment guidelines; To understand the different treatment options and its clinical outcomes, and to explore the best treatment options; To explore the best clinical pathway of PLC multidisciplinary consultation; To provide the basis for the development of clinical guidelines for PLC in China.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PLC after January 1,2012;
* First treatment and efficacy evaluation.

Exclusion Criteria:

* Complicated with another primary malignant tumor and secondary liver cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had been diagnosed with PLC were chosen
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2017-08-31 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival

IPD SHARING:
Plan to Share IPD: No